CLINICAL TRIAL: NCT00776035
Title: Sex and Obesity Effects on Myocardial Blood Flow and Metabolism
Brief Title: Sex and Obesity: Effects on Heart Failure Study
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 07-1128
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Heart Failure
Keywords: Obesity; Heart; Failure; PET (positron emission tomography); radiation; metabolism
MeSH Terms: conditions — Obesity; Heart Failure | interventions — Magnetic Resonance Spectroscopy; Caves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non diagnostic genetic samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Men with heart failure: Men with obesity-related heart failure
  Interventions: Procedure: PET (Positron Emission Tomography); Procedure: Echocardiogram; Radiation: ^15O-water; Radiation: 1-^11C-palmitate; Radiation: 1-^11C-glucose
- Women with heart failure: Women with obesity-related heart failure
  Interventions: Procedure: PET (Positron Emission Tomography); Procedure: Echocardiogram; Radiation: ^15O-water; Radiation: 1-^11C-palmitate; Radiation: 1-^11C-glucose

INTERVENTIONS:
Procedure: PET (Positron Emission Tomography) — This is a diagnostic scan that requires the injection of radioactive tracer compounds intravenously using an IV placed in the arm.
  Other Names: PET scan
Procedure: Echocardiogram — An echocardiogram is an ultrasound of the heart. Participants received a complete 2D- and Doppler echocardiographic examination on the day of the PET scan.
  Other Names: Echo
Radiation: ^15O-water — This is a radioactive tracer used to study blood flow in the heart during the PET scan. It was administered intravenously at a dose of 20 mCi.
Radiation: 1-^11C-palmitate — This is a radioactive tracer used to study fatty acid usage in the heart during the PET scan. It was administered intravenously at a dose of 20 mCi.
Radiation: 1-^11C-glucose — This is a radioactive tracer used to study glucose usage in the heart during the PET scan. It was administered intravenously at a dose of 20 Mci..

SUMMARY:
Sex has a major impact on myocardial metabolism and blood flow. In those without heart failure men's hearts tend to use proportionally more glucose and women's hearts use more fat and have higher blood flow.

Obesity is a major risk factor for Heart Failure. In those without heart failure, increasing body mass index is predictive of increased blood flow and fatty acid metabolism in women, but not men.

To measure blood flow and metabolism we used radioactive materials and a PET (positron emission Tomography) scan to study the blood flow and substrate metabolism of the heart.

Hypotheses: 1) Women with heart failure with reduced ejection fraction (HFrEF) will have higher levels of heart blood flow and fatty acid metabolism and lower glucose metabolism rates than men with HFrEF. A secondary Aim was to test the hypothesis that body mass index (BMI), a measure of obesity, correlated with myocardial blood flow and myocardial metabolism measures in patients with HFrEF.

ELIGIBILITY:
Inclusion criteria

* Heart failure (HF) and a systolic ejection fraction <45% per a recent echocardiogram report)
* Nonischemic HF New York Heart Association Class II-III
* Ambulatory
* Able to give informed consent
* On a stable medical regimen including the standard-of-care HF medications (i.e., a beta-blocker, ACE-inhibitor or angiotensin receptor blocker [ARB])

Exclusion criteria

* Participants who were pregnant or lactating
* Actively losing weight
* Nonsedentary (performing aerobic exercise > 30 minutes x 3 times/week)
* Those who have more than Class I hypertension
* Those who require alterations in beta-blocker or ACE or ARB-inhibition medication
* Those with hypertrophic, constrictive, or restrictive cardiomyopathies
* Those unable to lie flat in the PET scanner
* Severe major organ system dysfunction (other than heart failure)
* Significant coronary artery disease by catheterization
* Those unable to give informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males and females assigned so at birth are eligible to participate. Since the purpose was to evaluate sex-related differences in blood flow and metabolism without the effects of exogenous hormones, those taking the latter were excluded.
Study Population: Participants with heart failure were recruited for this study from the Washington University in St. Louis VO2 peak database, which consisted of participants who had been referred to and completed VO2 testing in the Cardiac Rehabilitation-run laboratory since 1998.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2000-02-01 (Actual); Primary Completion 2011-04-02 (Actual); Study Completion 2011-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Peterson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Essop MF, Opie LH. Metabolic therapy for heart failure. Eur Heart J. 2004 Oct;25(20):1765-8. doi: 10.1016/j.ehj.2004.08.019. No abstract available. PMID 15474689
- [Background] Taegtmeyer H, Salazar R. Myocardial metabolism: a new target for the treatment of heart disease? Curr Hypertens Rep. 2004 Dec;6(6):414-5. doi: 10.1007/s11906-004-0033-5. No abstract available. PMID 15527683
- [Background] Stanley WC, Recchia FA, Lopaschuk GD. Myocardial substrate metabolism in the normal and failing heart. Physiol Rev. 2005 Jul;85(3):1093-129. doi: 10.1152/physrev.00006.2004. PMID 15987803
- [Background] Kenchaiah S, Evans JC, Levy D, Wilson PW, Benjamin EJ, Larson MG, Kannel WB, Vasan RS. Obesity and the risk of heart failure. N Engl J Med. 2002 Aug 1;347(5):305-13. doi: 10.1056/NEJMoa020245. PMID 12151467
- [Background] Peterson LR, Herrero P, Schechtman KB, Racette SB, Waggoner AD, Kisrieva-Ware Z, Dence C, Klein S, Marsala J, Meyer T, Gropler RJ. Effect of obesity and insulin resistance on myocardial substrate metabolism and efficiency in young women. Circulation. 2004 May 11;109(18):2191-6. doi: 10.1161/01.CIR.0000127959.28627.F8. Epub 2004 May 3. PMID 15123530
- [Background] Kates AM, Herrero P, Dence C, Soto P, Srinivasan M, Delano DG, Ehsani A, Gropler RJ. Impact of aging on substrate metabolism by the human heart. J Am Coll Cardiol. 2003 Jan 15;41(2):293-9. doi: 10.1016/s0735-1097(02)02714-6. PMID 12535825
- [Background] Peterson LR, Soto PF, Herrero P, Schechtman KB, Dence C, Gropler RJ. Sex differences in myocardial oxygen and glucose metabolism. J Nucl Cardiol. 2007 Jul;14(4):573-81. doi: 10.1016/j.nuclcard.2007.03.001. Epub 2007 Jun 27. PMID 17679067
- [Background] Davila-Roman VG, Vedala G, Herrero P, de las Fuentes L, Rogers JG, Kelly DP, Gropler RJ. Altered myocardial fatty acid and glucose metabolism in idiopathic dilated cardiomyopathy. J Am Coll Cardiol. 2002 Jul 17;40(2):271-7. doi: 10.1016/s0735-1097(02)01967-8. PMID 12106931

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with nonischemic heart failure
Period: Overall Study
Arm/Group | Men With Heart Failure | Women With Heart Failure
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants with nonischemic heart failure
Groups:
- Total: Total of all reporting groups
Arm/Group | Men With Heart Failure | Women With Heart Failure | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (3) | 41 (3) | 41.5 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 10 | 10
  Male | 9 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Homeostasis model assessment of insulin resistance [Mean (Standard Deviation); unit: units on a scale] — HOMA-IR is a method to estimate insulin resistance. It is calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5. A score of <1 indicates insulin-sensitivity; >1.9 indicates early insulin resistance; and >2.9 indicates significant insulin resistance.
  units on a scale | 2.55 (0.51) | 4.40 (1.77) | 3.52 (4.19)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is a measure of body fat based on height and weight. It is calculated as body weight divided by the square of body height. Underweight = <18.5; normal weight = 18.5 to 24.9; overweight = 25 to 29.9; and obesity is >30.
  kg/m^2 | 31 (2) | 35 (8) | 32.96 (7.54)

OUTCOME MEASURES:

1. Primary Outcome: Average Myocardial Blood Flow
Description: Myocardial blood flow (MBF) was measured using ^15O-water injected intravenously intravenously through a large bore catheter into an antecubital vein during the (Positron Emission Tomography (PET) scan on Study Day 2.
Time Frame: Study Day 2
Population: Participants who completed the PET scan assessment
Measure: Mean (Standard Deviation); unit: mL/g/minute
Arm/Group | Men With Heart Failure | Women With Heart Failure
Number analyzed (Participants) | 9 | 10
mL/g/minute | 0.73 (0.17) | 0.97 (0.13)
Statistical Analysis 1: Comparison: Men With Heart Failure vs Women With Heart Failure; Average myocardial blood flow, men versus women; Test type: Superiority; p < 0.005, Student's t-test

2. Secondary Outcome: Average Myocardial Fatty Acid Utilization
Description: Myocardial fatty acid (FA) utilization was measured using 1-^11C-palmitate injected intravenously through a large bore catheter into an antecubital vein during the (Positron Emission Tomography (PET) scan on Study Day 2.
Time Frame: Study Day 2
Population: Participants who completed the PET assessment
Measure: Mean (Standard Deviation); unit: nmol/g/minute
Arm/Group | Men With Heart Failure | Women With Heart Failure
Number analyzed (Participants) | 9 | 10
nmol/g/minute | 85 (26) | 139 (68)
Statistical Analysis 1: Comparison: Men With Heart Failure vs Women With Heart Failure; Average myocardial fatty acid utilization, men versus women; Test type: Superiority; p < 0.05, Student's t-test

ADVERSE EVENTS:
Time Frame: All-cause mortality and treatment-emergent adverse events were collected from Study Day 1 to 48 hours after Study Day 2.
Arm/Group | Men With Heart Failure | Women With Heart Failure
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes